CLINICAL TRIAL: NCT05414461
Title: Efficacy of PD-1-inhibitor-based Combination Therapy in Patients With Metastatic Colorectal Cancer
Brief Title: Efficacy of Combination Immunotherapy in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Feng Ye, Chief physician, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CombiImmuno mCRC
Record Dates: First submitted 2022-06-04; First posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination treatment (Experimental): PD-1 inhibitor-based combination treatment
  Interventions: Drug: Combinations

INTERVENTIONS:
Drug: Combinations — PD-1 inhibitor-based combinaiton treatment

SUMMARY:
Immunotherapy improved efficacy and survival in selective patients with metastatic colorectal cancer (mCRC), however, limited data revealed the landscape of immunotherapy efficacy. What's more, potential markers have not been comprehensively evaluated to identify responding patients to further improve efficacy.The investigators conducted a single-arm study to investigate the efficacy of combination immunotherapy in patients with mCRC, and the combined regimen is determined by the physician in charge.

ELIGIBILITY:
Inclusion Criteria:

* patients who had both baseline measurable lesion(s) and at least one post-baseline radiological disease reassessment
* patients with identified genomic status

Exclusion Criteria:

* patients who received immune monotherapy
* patients who stopped treatment for any reason without identified response assessment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2021-10-17 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Durable clinical benefit | immediately after the intervention
  Rate of patients who acheived CR or PR or SD that lasted more than 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No